CLINICAL TRIAL: NCT02321657
Title: RELAX Anaesthetics: the Effect of a Bespoke Relaxation App on Stress Levels in Children Undergoing Anaesthesia
Acronym: RELAX-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Music (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RELAX2015
Record Dates: First submitted 2014-12-08; First posted 2014-12-22 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iPad app containing art, music and games (Experimental): On entry to the anaesthetic room, children will be given an iPad (the intervention) with art, music and games to distract them. A nurse will help them engage with the iPad whilst the anaesthetists complete the anaesthetic. Once the child falls asleep, the iPad will be removed. This process is anticipated to last between 3 and 30 minutes depending on the time taken to anaesthetise the child.
  Interventions: Other: iPad app containing art, music and games
- Toys, books and games (Active Comparator): On entry to the anaesthetic room, children will be given toys or games to distract them. A nurse will help them play whilst the anaesthetists complete the anaesthetic. Once the child falls asleep, the games will be removed. This process is anticipated to last between 3 and 30 minutes depending on the time taken to anaesthetise the child.
  Interventions: Other: Toys, books and games

INTERVENTIONS:
Other: iPad app containing art, music and games — An iPad app that takes demographic information on a child and suggests suitable art, music and games for use by the anaesthetist and nurse to distract them during anaesthetics
  Arms: iPad app containing art, music and games
Other: Toys, books and games — Games, books and toys used to distract
  Arms: Toys, books and games

SUMMARY:
RELAX Anaesthetics is a randomised clinical trial assessing the effectiveness of using an iPad app with art, music and games to relax and distract children, reduce anaesthetic induction time and make drug cost savings prior to surgery.

DETAILED DESCRIPTION:
The most distressing part of a parent's experience in hospital is watching a child undergo intravenous cannulation.1 This is commonly performed in the anaesthetic room prior to induction of anaesthesia. At Chelsea and Westminster Foundation Trust (CWFT) over 5000 children undergo operations every year. Traditional methods of distracting the child during have included blowing bubbles, storybooks, and a variety of toys and games. These methods are not always effective and may present an infection risk due to inability to clean between uses.

The use of an android/iPad provides a platform for effectively distracting the child with a choice of games, video and music, with the advantage of being cleaned between uses. Users of this platform are required to select the application that is most appropriate for the age, sex, method of anaesthesia, and compliance level of the child. To assist with this, the investigators have developed an application system that will select a range of entertainment applications appropriate for each child based on these four variables and hopefully help to keep children calm before their operations.

ELIGIBILITY:
Inclusion Criteria:

* children ages 2 -12 years
* requiring general anaesthesia
* ASA assessment of fitness for surgery score 1 - 3

Exclusion Criteria:

* intravenous cannula already in situ
* play therapist already in use
* anaesthetist refusal to participate
* parental / patient refusal to participate
* sedative or opiate pre-med already administered
* not requiring general anaesthesia
* ASA assessment of fitness for surgery score 4 or 5

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale | Change between baseline and completion of cannulation (2 hours later)
  An observational scale assessing distress levels

SECONDARY OUTCOMES:
Paediatric Anaesthetic Emergence Delirium Score | Single measurement taken from observation over 15 minutes immediately following surgery
  An observational scale assessing delirium levels post surgery
State Trait Anxiety Inventory | Change between baseline and completion of cannulation (2 hours later)
  A psychological scale measuring parental anxiety before and following the anaesthetic procedure for their child

OTHER OUTCOMES:
Time to induction | Duration of anaesthetics timed (from entering the anaesthetics room to successful anaesthetisation of child (estimated 3-30mins in the room)
  Time taken to cannulate and anaesthetise a child
Drugs cost | Drugs used from the time the child enters the anaesthetics room to successful anaesthetisation (estimated 3-30mins in the room)
  Cost of induction agents during anaesthetic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brooks, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital, London
  - Centre for Performance Science, Royal College of Music, London